CLINICAL TRIAL: NCT03525275
Title: The Effect of Battlefield Acupuncture and Physical Therapy Versus Physical Therapy Alone Following Shoulder Surgery: A Randomized Clinical Trial
Brief Title: Effect of Battlefield Acupuncture and Physical Therapy Versus Physical Therapy Alone After Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Keith Collinsworth, Principle Investigator, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USMA BFA
Record Dates: First submitted 2018-04-27; First posted 2018-05-15 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Opioid Use; Pain, Postoperative; SLAP Lesion; Bankart Lesion; Subacromial Impingement Syndrome; Rotator Cuff Tear; Glenohumeral Dislocation; Glenohumeral Subluxation; Hill Sach Lesion; Bony Bankart Lesion; Acromioclavicular Separation
MeSH Terms: conditions — Pain, Postoperative; Bankart Lesions; Shoulder Impingement Syndrome; Rotator Cuff Injuries; Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: 2 x 5 Mixed model ANOVA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFA with Physical Therapy (Experimental): BFA + post-surgical protocol, intervention = battlefield acupuncture plus post-surgical protocol
  Interventions: Device: Battlefield Acupuncture; Procedure: Post-surgical shoulder protocol
- Physical Therapy alone (Active Comparator): Intervention = Post-surgical protocol
  Interventions: Procedure: Post-surgical shoulder protocol

INTERVENTIONS:
Device: Battlefield Acupuncture — Battlefield Acupuncture uses ASP semi-permanent needles inserted into their ears for pain attenuation in 5 known points. Both groups receive their respective post-surgical rehabilitation protocols
  Arms: BFA with Physical Therapy
Procedure: Post-surgical shoulder protocol — Surgery specific post-surgical physical therapy protocol

SUMMARY:
The purpose of this randomized clinical trial is to determine the effectiveness of Battlefield Acupuncture (BFA) in addition to usual post-surgical shoulder physical therapy compared to a standard shoulder rehabilitation program in reducing medication use and pain in patients who have undergone shoulder surgery. Measurements of medication (opioid, NSAID, acetaminophen, etc.) use (daily number of pills consumed), pain rating, patient specific functional scale and global rating of change will be taken at 24, 72 hours, 7 days, 14 days and at six weeks post-surgery. It is hypothesized that the inclusion of Battlefield Acupuncture will result in a decrease in medication use and post-surgical pain when compared to rehabilitation alone. The population for this study is male and female DoD beneficiaries, ages 17-55 (17 if cadet) that are not participating in other shoulder research studies. The subjects in the experimental group will receive Battlefield Acupuncture in addition to their respective post-surgical shoulder rehabilitation protocol.

DETAILED DESCRIPTION:
GROUPS Group assignment will be recorded with individual subject identifier and secured in a separate folder until completion of all data collection through the final follow up.

* Experimental Group: Battlefield Acupuncture with respective shoulder surgery protocol
* Control Group: respective post-surgical Shoulder protocol

All Battlefield Acupuncture will be performed by the PI or AI's who are trained in Battlefield Acupuncture. The Battlefield Acupuncture technique will be standardized. The subject will continue to receive the standard of care in accordance with the post-operative protocol between follow-ups.

Experimental Group: Subjects in the experimental group will receive the usual post-surgical rehabilitation protocol per their surgery in addition to Battlefield Acupuncture. Using sterile technique, Battlefield acupuncture using the 5 points within the Battlefield Acupuncture protocol will be used until the desired 0-1/10 VAS is reported by the subject. The sequencing of the acupuncture begins on the same side of the shoulder surgery. Each ear has 5 points of puncture by the ASP needles. The points, in sequence of puncture are named: cingulate gyrus, thalamus, omega 2, point zero and shen men. The PA/AI using sterile technique (proper hand washing, PPE) will start with the ipsilateral ear. The subjects ear is cleaned with an alcohol swab, and punctured with the ASP needle in the cingulate gyrus. After waiting for pain attenuation/side effect monitoring, the subject will ambulate in the clinic to reassess their perceived pain. If the subjects' pain is above the desired 0-1/10 VAS level, the contralateral ear will be punctured with the ASP needle in the cingulate gyrus under sterile technique. After waiting for pain attenuation/side effect monitoring, the subject will ambulate in the clinic to reassess their perceived pain. If the subjects' pain is above the desired 0-1/10 VAS level, the ipsilateral ear will be punctured with the ASP needle in the thalamus point under sterile technique. After waiting for pain attenuation/side effect monitoring, the subject will ambulate in the clinic to reassess their perceived pain. This sterile acupuncture process will proceed alternating ears until the dominant ear for pain attenuation is determined (using only the 5 Battlefield Acupuncture points) until the desired 0-1/10 VAS level is achieved. The subject will be constantly monitored for side effects to include light headedness, dizziness/loss of balance or nausea. Depending on the subjects' pain response, the ASP needles may be inserted into one ear predominantly, for greater pain attenuation. The ASP needles may remain in the Subjects' ears for 3-5 days. There is no standard time for the ASP needles to remain in the Subjects' ears. The ASP needles will naturally work their way out of the Subject's skin over 3-5 days. There are no documented cases of loss of treatment effect if the Subject removes the ASP needles premature to their natural falling off.

Control Group: Subjects in this group will receive rehabilitation and will perform a home exercise program in accordance with the post-operative shoulder protocol. Subjects will be asked to record compliance on an exercise log. Handouts will be provided to each subject.

Repeat measurement of VAS, PSFS, GROC, and daily opioid/NSAID/acetaminophen use will be taken by the PI/AI or study staff on day one, 72 hours, 7days, 14 days and at 6weeks.

All study subjects will engage in supervised progression of their respective post-surgical protocols. Subjects will be progressed within their respective protocols at a safe pace, and their home exercise program compliance will be monitored throughout the 6 weeks of this study. At any time, a subject may opt out of the study without detriment in their care at KACH/Arvin Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Department of Defense beneficiaries ages 17-55, prior to or recent (within 24 hrs) shoulder surgery

Exclusion Criteria:

* Self-reported pregnancy, History of blood borne pathogens/infectious disease/active infection/metal allergy, bleeding disorders or currently taking anti-coagulant medications, Participants who are not fluent in English

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain medication use | daily log, comparison at 24hours, 72hours, 1 week, 2 weeks, 6 weeks
  Patient log of daily pain medication use (opioid, NSAID, acetaminophen), the number of pills per medication will be logged daily over the course of 6 weeks
Change in Visual Analog Pain scale report | outcome comparison at 24hours, 72hours, 1 week, 2 weeks, 6 weeks
  patient's perceived pain on the Visual Analog Scale, 0 to 100mm scale with higher equaling more pain perceived by the subject, 0 = no pain and 10= worst pain imaginable.

SECONDARY OUTCOMES:
Change in Global Rating of Change (GROC) | outcome comparison at 24 hours, 72hours, 1 week, 2 weeks, 6 weeks
  Patient perceived improvement from time of surgery using Global Rating of Change, Scored [-7 to 0 to +7] with 0= "no change", -7 "= "a very great deal worse" and +7="a very great deal better".
Change in Patient Specific Functional Scale (PSFS) | outcome comparison at 24 hours, 72hours, 1 week, 2 weeks, 6 weeks
  Patient perceived functional difficulty in self selected tasks, 0 to 10 scale with 0= unable to perform specific activity and 10 = "able to perform activity the same as prior to surgery".

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Collinsworth, DPT, Principal Investigator — Keller ACH
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No